CLINICAL TRIAL: NCT01512823
Title: Randomised Trial of the Effectiveness of Two Educational Interventions to Improve Evidence-based Practice Knowledge, Attitudes and Behaviour in Occupational Therapists
Brief Title: Randomised Trial of Two Educational Intervention for Improving Evidence-based Practice Knowledge, Atttitudes and Practice
Acronym: OTEBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cape Town (Other)
Collaborators: National Research Foundation of South Africa (Other)
Responsible Party: Principal Investigator, Helen Buchanan, Principal investigator, University of Cape Town
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: REC REF: 259/2006
Record Dates: First submitted 2012-01-13; First posted 2012-01-19 (Estimated); Last update posted 2012-02-06 (Estimated); Status verified 2012-02

CONDITIONS: Health Knowledge, Attitudes, Practice
Keywords: randomised controlled trial; educational intervention; occupational therapy
MeSH Terms: conditions — Behavior | interventions — Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interactive educational intervention (Experimental): Two education sessions (four-hours and two-hours respectively), emailed notes and reminders
  Interventions: Behavioral: Education
- Didactic educational intervention (Experimental): Education alone
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Education — Interactive educational intervention:
  * 4 hour education session (with notes and 'evidence packs'); presentations, small group discussion tasks and practice of particular skills - 2 hour session (1 week later)
  * Emailed notes from second session
  * Telephonic/email follow-up (reminders)
  Didactic educational intervention:
  - 4 hour education session (with notes and 'evidence packs'; questions answered but no discussion or application of skills

SUMMARY:
This pragmatic randomised controlled trial (RCT) used a two-group parallel design with matched-pair stratification by type (clinician/manager) and knowledge score. The trial aimed to: 1) determine whether an IE was more effective than a DE for improving EBP knowledge, skills and use at 12 weeks, and 2) to investigate the feasibility of conducting a RCT with occupational therapists in a public health setting. Occupational therapists employed by the Western Cape Department of Health (DOH) form,ed the study population(N=98). Fifty-eight consented to participate and were randomly allocated to either an interactive (IE) or a didactic (DE) educational intervention using coin tossing. Data was collected at baseline and 12 weeks The primary outcome was increased EBP knowledge at 12 weeks shown by an improved total knowledge score. Secondary outcomes were improved attitudes and behaviour. Data were collected at the health facilities where participants were employed. Raters for the audit were blinded but participants and the provider could not be blinded.

Thirty participants were allocated to receive the IE and 28 the DE. Twenty-five participants in the IE and 21 in the DE completed the trial and were included in the 12 week analysis. Results revealed no significant difference between the groups in the primary knowledge outcome at 12 weeks. Examination of within-group changes revealed significant improvements in knowledge in both groups (IE: T=4.0, p<0.001; DE: T=12.0, p=0.002), but the IE also showed a significant increase in behaviour (T=64.5, p=0.044) and attitudes on one sub-scale (T=33.0, p=0.039). As the study was powered at 43%, it may have failed to detect significant differences at 12 weeks. Conducting a high-quality RCT was feasible and the risk of bias was assessed as low. The OTEBP trial adds strength to the existing evidence that both didactic and interactive educational interventions can improve knowledge, but it seems that interactive interventions may be more effective for changing behaviour. High-quality pragmatic trials can feasibly be conducted within the public health service

ELIGIBILITY:
Inclusion Criteria:

* Occupational therapists employed by the Western Cape Department of Health (DOH)
* Working at least 20 hours per week

Exclusion Criteria:

* Working at a distance of more than 1½ hours from Cape Town
* Therapists who would be leaving the DOH before December 2008 or taking leave during the time of the intervention

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2007-11; Primary Completion 2009-01 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Shortened Fresno Test of Competence in Evidence-based Practice (SAFT) | 12 weeks
  Modified from the Adapted Fresno Test of Competence in EBP (AFT) (McCluskey and Bishop, 2009), the SAFT consists of three items testing knowledge of writing a PICO question based on a clinical scenario, ability to identify the most suitable study design to answer the question, and knowledge of possible sources of information. The total possible score is 30 points. The test is scored using a grading rubric. Two versions are availbale for measuring outcomes of educational interventions.

SECONDARY OUTCOMES:
Audit checklist | 12 weeks
  9-item checklist for auditing patient records to determine the extent to which occupational therapists monitor the effectiveness of their interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Helen Buchanan, PhD, Principal Investigator — University of Cape Town; Nandi Siegfried, PhD, Study Director — South African Cochrane Centre & University of Cape Town; Jennifer Jelsma, PhD, Study Director — University of Cape Town
Locations (1):
- University of Cape Town, Cape Town, Western Cape, South Africa

REFERENCES:
- [Derived] Buchanan H, Jelsma J, Siegfried N. Measuring evidence-based practice knowledge and skills in occupational therapy--a brief instrument. BMC Med Educ. 2015 Oct 30;15:191. doi: 10.1186/s12909-015-0475-2. PMID 26519165
- [Derived] Buchanan H, Siegfried N, Jelsma J, Lombard C. Comparison of an interactive with a didactic educational intervention for improving the evidence-based practice knowledge of occupational therapists in the public health sector in South Africa: a randomised controlled trial. Trials. 2014 Jun 10;15:216. doi: 10.1186/1745-6215-15-216. PMID 24916176